CLINICAL TRIAL: NCT02369172
Title: A Single-centre, Open-label Study in Healthy Men to Investigate the Effect of Repeated Oral Doses of ASP2151 on the Pharmacokinetics of Bupropion
Brief Title: Drug-Drug Interaction Study: ASP2151 and Bupropion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maruho Europe Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M522101-EU25
Record Dates: First submitted 2015-02-16; First posted 2015-02-23 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-01

CONDITIONS: Healthy
Keywords: Herpes; volunteers; drug-drug interaction
MeSH Terms: conditions — Herpes Simplex | interventions — Bupropion; ASP2151

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupropion + ASP2151 (Other): 400 mg ASP2151 followed by 150 mg Bupropion
  Interventions: Drug: Bupropion; Drug: ASP2151

INTERVENTIONS:
Drug: Bupropion
  Other Names: Zyban
Drug: ASP2151

SUMMARY:
CYP2B6 is involved in the metabolism of many drugs. So, it is important to assess in vivo the effect of ASP2151 on that enzyme to determine any possible drug interactions. The aim of this trial is to investigate the potential for interaction of ASP2151 with the CYP2B6 probe substrate bupropion.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (Quetelet index) in the range 18.0-30.9.
* Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
* Willingness to give written consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or his delegate.
* Willingness to give written consent to have data entered into The Overvolunteering Prevention System.

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
* Any of the following liver function tests higher than 1.5 times the ULN at the screening visit: aspartate aminotransferase (AST), alanine aminotransferase (ALT), ALP, bilirubin, gamma glutamyl transpeptidase (gamma-GT).
* Platelet counts outside normal limits (129,000-346,000/μL).
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
* Clinically significant impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
* History of bleeding diathesis, head injury, intracranial mass lesions, hydrocephalus, epilepsy, seizures, depression, self-harm (or thoughts of self-harm) or eating disorders.
* Surgery (eg stomach bypass) or medical condition that might affect absorption of medicines.
* Presence or history of severe adverse reaction to any drug, history of multiple drug allergies (multiple defined as >3), or sensitivity to trial medication.
* Use, during the 28 days before the first dose of trial medication, of any prescription medicine, or any other medicine or herbal remedy (such as St John's wort) known to interfere with the CYP3A4, CYP2C8, CYP2B6, CYP2D6 or CYP2C19 metabolic pathway.
* Use, during the 7 days before the first dose of trial medication, of any over-the-counter medicine, with the exception of paracetamol (acetaminophen).
* Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months.
* Presence or history of drug or alcohol abuse, or intake of more than 21 units of alcohol weekly.
* Current smoker or history of regular use of tobacco or nicotine-containing products within the previous 6 months.
* Blood pressure and heart rate in seated position at the screening examination outside the ranges 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40_100 beats/min. However, if the investigator deems the result to be not clinically significant the subject may be included.
* Possibility that the volunteer will not cooperate with the requirements of the protocol.
* Evidence of drug abuse on urine testing.
* Positive test for hepatitis B, hepatitis C, HIV1 or HIV2.
* Loss of more than 400 mL blood during the 3 months before the trial, eg as a blood donor.
* Objection by General Practitioner (GP) to volunteer entering trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research Ltd, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in United Kingdom from 03-February 2015 to 17-April 2015
Groups:
- Bupropion + ASP2151: 400 mg ASP2151 followed by 150 mg Bupropion
  Bupropion
  ASP2151
Period: Overall Study
Arm/Group | Bupropion + ASP2151
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bupropion + ASP2151
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 32.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 18
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax) of Bupropion
Time Frame: prior to initial dose of Day 1 and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 60, 72 and 96 h after dosing on Day 1, Days 15, 22 and 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Day 1; Day 22; Day 29: 150 mg bupropion alone
- Day 15: 150 mg bupropion with 400 mg ASP2151
Arm/Group | Day 1 | Day 15 | Day 22 | Day 29
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 91.28 (27.2) | 76.94 (30.3) | 92.21 (28) | 95 (25.2)

2. Primary Outcome: Area Under the Concentration-time Curve Extrapolated to Infinite Time (AUC0-∞) of Bupropion
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 1 | Day 15 | Day 22 | Day 29
Number analyzed (Participants) | 24 | 24 | 24 | 24
h*ng/mL | 777.6 (30) | 653.7 (26.1) | 785.5 (31.1) | 841.4 (29)

3. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Refer to the result of adverse event.
Time Frame: Up to 32 days after the last dose
Measure: Number; unit: participants
Groups:
- All Subjects: All subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 24
participants
  Non-serious adverse event | 12
  serious adverse event | 0

4. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of Hydroxybupropion
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Day 1 | Day 15 | Day 22 | Day 29
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 295.4 (30.9) | 300.7 (32.6) | 300.6 (27.5) | 291.6 (31.2)

5. Other Pre Specified Outcome: Time of Peak Concentration (Tmax) of Hydroxybupropion
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Day 1 | Day 15 | Day 22 | Day 29
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 8 [4.00 to 10.08] | 8 [5.00 to 24.00] | 8 [5.00 to 12.00] | 8 [3.00 to 12.02]

6. Other Pre Specified Outcome: Area Under Concentration-Time Curve up to Last Non-zero Value (AUC0-tn) of Hydroxybupropion
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 1 | Day 15 | Day 22 | Day 29
Number analyzed (Participants) | 24 | 24 | 24 | 24
h*ng/mL | 10524.7 (32.9) | 10160.7 (37.7) | 11135.4 (34.1) | 10963 (37.4)

7. Other Pre Specified Outcome: Area Under the Concentration-time Curve Extrapolated to Infinite Time (AUC0-∞) of Hydroxybupropion
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 1 | Day 15 | Day 22 | Day 29
Number analyzed (Participants) | 24 | 24 | 24 | 24
h*ng/mL | 11195.7 (33.7) | 10838.3 (38) | 12037.2 (36.1) | 11825.3 (38)

8. Other Pre Specified Outcome: Half-life (t1/2) of Hydroxybupropion
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Day 1 | Day 15 | Day 22 | Day 29
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 21.38 (20.6) | 20.97 (20.3) | 23.07 (23.8) | 22.89 (16.8)

9. Other Pre Specified Outcome: Trough Plasma Concentration (Ctrough) of ASP2151
Time Frame: Days 6-14 and at pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h after dosing on Day 15
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Day 6: Day 6 pre-dose
- Day 7: Day 7 pre-dose
- Day 8: Day 8 pre-dose
- Day 9: Day 9 pre-dose
- Day 10: Day 10 pre-dose
- Day 11: Day 11 pre-dose
- Day 12: Day 12 pre-dose
- Day 13: Day 13 pre-dose
- Day 14: Day 14 pre-dose
- Day 15: Day 15 pre-dose
Arm/Group | Day 6 | Day 7 | Day 8 | Day 9 | Day 10 | Day 11 | Day 12 | Day 13 | Day 14 | Day 15
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
ng/mL | 0 (0) | 244.95 (104.63) | 245.83 (122.39) | 219.17 (105.83) | 185.31 (84.66) | 199.16 (105.72) | 197.05 (99.95) | 192.66 (102.29) | 188.46 (95.75) | 178.93 (87.78)

10. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of ASP2151
Time Frame: prior to initial dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h after dosing on Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Day 15
Number analyzed (Participants) | 24
ng/mL | 1409.8 (33.7)

11. Other Pre Specified Outcome: Time of Peak Concentration (Tmax) of ASP2151
Time Frame: prior to initial dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h after dosing on Day 15
Measure: Median (Full Range); unit: h
Arm/Group | Day 15
Number analyzed (Participants) | 24
h | 3 [1.00 to 5.00]

12. Other Pre Specified Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUC0-tau) of ASP2151
Time Frame: prior to initial dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h after dosing on Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 15
Number analyzed (Participants) | 24
h*ng/mL | 14201.4 (33.5)

13. Other Pre Specified Outcome: Area Under the Concentration-time Curve Extrapolated to Infinite Time (AUC0-∞) of ASP2151
Time Frame: prior to initial dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h after dosing on Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 15
Number analyzed (Participants) | 24
h*ng/mL | 15968.1 (35.1)

14. Other Pre Specified Outcome: Half-life (t1/2) of ASP2151
Time Frame: prior to initial dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h after dosing on Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Day 15
Number analyzed (Participants) | 24
h | 7.198 (16.7)

15. Other Pre Specified Outcome: Apparent Volume of Distribution (Vd/F) of ASP2151
Time Frame: prior to initial dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h after dosing on Day 15
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Day 15
Number analyzed (Participants) | 24
L | 274 (97.85)

16. Other Pre Specified Outcome: Apparent Total Body Clearance (CL/F) of ASP2151
Time Frame: prior to initial dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h after dosing on Day 15
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Day 15
Number analyzed (Participants) | 24
L/h | 26.43 (8.65)

17. Other Pre Specified Outcome: Time of Peak Concentration (Tmax) of Bupropion
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Day 1 | Day 15 | Day 22 | Day 29
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 3 [2.00 to 6.00] | 3 [1.00 to 5.98] | 3 [2.00 to 5.00] | 3 [1.00 to 5.00]

18. Other Pre Specified Outcome: Area Under the Curve Over up to Last No-zero Value (AUC0-tn) of Bupropion
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 1 | Day 15 | Day 22 | Day 29
Number analyzed (Participants) | 24 | 24 | 24 | 24
h*ng/mL | 732.3 (29.9) | 608.9 (26.5) | 742.8 (31.8) | 794.2 (29.4)

19. Other Pre Specified Outcome: Half-life (t1/2) of Bupropion
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Day 1 | Day 15 | Day 22 | Day 29
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 9.76 (47.7) | 8.16 (42.1) | 9.13 (37) | 10.92 (42.7)

20. Other Pre Specified Outcome: Apparent Volume of Distribution (Vd/F) of Bupropion
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Day 1 | Day 15 | Day 22 | Day 29
Number analyzed (Participants) | 24 | 24 | 24 | 24
L | 2801.5 (723.1) | 2791.4 (747.05) | 2581.2 (588.69) | 2979.7 (1124.63)

21. Other Pre Specified Outcome: Apparent Total Body Clearance (CL/F) of Bupropion
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Day 1 | Day 15 | Day 22 | Day 29
Number analyzed (Participants) | 24 | 24 | 24 | 24
L/h | 200.64 (56.33) | 236.46 (57.2) | 199.59 (62.04) | 185.59 (57.71)

ADVERSE EVENTS:
Time Frame: Up to 32 days after the last dose
Groups:
- Bupropion: after dosing with bupropion on Day 1 and before the first dose of ASP2151 on Day 6.
- ASP2151 After Bupropion: after the first dose of ASP2151 on Day 6, and before co-administration of bupropion and ASP2151 on Day 15.
- Bupropion With ASP2151: after co-administration of bupropion and ASP2151 on Day 15.
Arm/Group | Bupropion | ASP2151 After Bupropion | Bupropion With ASP2151 | Total
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/24 | 5/24 | 10/24 | 12/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion (N=24) | ASP2151 After Bupropion (N=24) | Bupropion With ASP2151 (N=24) | Total (N=24)
Headache (Nervous system disorders) | 1 | 2 | 4 | 6
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1
Catheter site pain (General disorders) | 0 | 1 | 1 | 2
Catheter site haematoma (General disorders) | 0 | 0 | 1 | 1
Catheter site phlebitis (General disorders) | 0 | 0 | 1 | 1
Catheter site related reactions (General disorders) | 1 | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 2 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1
Abdominal (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Concstipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No